CLINICAL TRIAL: NCT04774874
Title: A Randomized, Double-blind, Vehicle-controlled, Dose-finding Multi-center, Phase 2a Trial of FOL-005 Topical Formulations to Investigate Hair Growth Potential and Safety in Healthy Male Volunteers With Androgenetic Alopecia
Brief Title: A Phase 2a Trial of FOL-005 Topical Formulations to Investigate Hair Growth Potential and Safety in Healthy Male Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Follicum AB (Industry)
Collaborators: proDERM GmbH (Industry); Hair and Skin Institute, Charité, Berlin, Germany (Unknown); CentroDerm GmbH (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCS-003
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial will be conducted as a double-blind trial. Neither the Investigator nor the subject will know the identity of the IP assigned. Also, all other persons involved in the trial (e.g. Data Manager and Trial Statistician) remain blinded until all possible queries are resolved and 'closure of the data base' is done, i.e. after quality assurance of the data and hard lock of the data base clean files.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- FOL- 005 (0.1 %) (Experimental): topical formulation
  Interventions: Drug: Topical formulation
- FOL -005 (0.5 %) (Experimental): topical formulation
  Interventions: Drug: Topical formulation
- FOL -005 (1.5 %) (Experimental): topical formulation
  Interventions: Drug: Topical formulation
- Vehicle (Placebo Comparator): topical formulation
  Interventions: Drug: Topical formulation

INTERVENTIONS:
Drug: Topical formulation — Topical administration on the scalp once daily for 16 weeks

SUMMARY:
This exploratory phase IIa, double blind, randomized, vehicle controlled, multicenter dose-finding trial will evaluate the safety, tolerability, and efficacy of FOL-005 topical formulation (at 0.1%, 0.5% and 1.5% strength) administered once daily (in the evening) for 16 weeks in healthy male subjects with androgenetic alopecia.

DETAILED DESCRIPTION:
This exploratory phase IIa, double blind, randomized, vehicle controlled, multicenter dose-finding trial will evaluate the safety, tolerability, and efficacy of FOL-005 topical formulation (at 0.1%, 0.5% and 1.5% strength) administered once daily (in the evening) for 16 weeks in healthy male subjects with androgenetic alopecia.

The trial will be performed at three centers in Germany. The aim of the trial is to determine the most efficacious dose of FOL-005 topical formulation based on efficacy dose trends. It is planned to randomize 220 subjects (with a ratio 1:1:1:1 FOL-005 0.1%; FOL-005 0.5%; FOL-005 1.5%; vehicle).

The trial consists of a screening period of up to three weeks and a treatment period of 16 weeks.

Eligible subjects will be randomized at Baseline (Day 1) and will apply the investigational products themselves at home once daily for 16 weeks. Subjects will return to the sites bi- weekly for check of compliance and assessment of local tolerability. At Day1, Day 84 and Day 112 subjects will be evaluated for hair growth parameters by TrichoLAB imaging. The end of the clinical trial for each individual subject is defined as the Final Visit at Day 112. In case of premature termination of a randomized subject an Early Termination (ET) visit should be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male, aged 18-55 years
2. Skin phototype II, III and IV according to Fitzpatrick's classification (Fitzpatrick et al. 1974)
3. Androgenetic alopecia (AGA) classified according to Hamilton Norwood grade 3V, 4, 5, 5A, 5V (Hamilton, 1951)
4. Willing and able to comply with scheduled visits
5. Willing to maintain the same hair hygiene products and general hair care habits during the trial period
6. Willing to maintain the same hair length and hair color during the trial period
7. Willing to have treatment areas shaved for TrichoLAB® measurement and marked with small semi-permanent dot tattoos
8. Willing to avoid prolonged UV exposition and UV tanning beds
9. Signed written informed consent before participation in the trial.
10. Subjects with a hair length of above 1 cm

Exclusion Criteria:

1. Damaged skin in or around test sites including sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test sites risking to interfere with investigational evaluations
2. Any dermatological disorders of the scalp which might interfere with the application of the investigational product (IP) or examination method, such as fungal or bacterial infections, seborrheic dermatitis (except mild forms which are managed with OTC shampoos and which do not require dermatological treatment), psoriasis, eczema, folliculitis, that require chronic use of medication or scalp atrophy
3. Any skin pathology (e.g. scar, nevus) or general condition (e.g. uncontrolled thyroid diseases) that in the Investigator's opinion can interfere with the evaluation of the test areas or requires prohibited topical or systemic therapy
4. History of active hair loss due to alopecia areata, scarring alopecia, diffuse telogen effluvium or conditions other than androgenetic alopecia
5. Diabetes mellitus
6. Presence of any acute (e.g. acute infections) or chronic illness (e.g. psoriasis, atopic dermatitis, porphyria, folliculitis) or presence or history of known skin cancer that in the opinion of the Investigators might confound the results of the trial
7. History or clinical signs of keloids or hypertrophic scars
8. Immunological disorders such as alopecia areata, and systemic lupus erythematosus and other systemic known autoimmune disorders
9. Current or within the last 6 months history of severe dietary or weight changes
10. Hair transplantation at any time
11. Known sensitization to cosmetic hair dyes or hypersensitivity to any ingredients of the IP or tattoo ink.
12. Application of topical minoxidil preparation or any other topical over-the counter (OTC) or prescription medication for hair re-growth to scalp for 4 weeks or more during a 6 months period before enrollment.
13. Use of or planned use of shampoo with expected medicinal effect on the scalp (e.g. but not limited to anti-dandruff containing ketoconazole, anti-psoriatic, anti-fungal or shampoo containing urea, caffeine, acetylsalicylic acid, etc.) during the course of trial
14. Topical treatments of the scalp including corticosteroids, tacrolimus, retinoids or other treatments that may affect hair growth in the last 3 months as well as during the trial.
15. Platelet rich plasma (PRP) or any mesotherapy treatment on scalp during the last 12 months as well as during the trial.
16. Systemic therapy using retinoids, cyclosporine, beta blockers or corticosteroids within the last 6 months as well as during the trial.
17. Scalp procedures e.g. surgery, laser, light, micro-needling within the last 6 months as well as during the trial.
18. Finasterid (e.g. Propecia®) or Dutasteride intake or topical application in the last 12 months, or any systemic hair therapy medication in the last 12 months as well as during the trial.
19. Other systemic therapy which in the opinion of the Investigator might affect hair growth
20. Current or within 2 weeks prior to first dosing use of vasodilating drugs (e.g. Pentoxifyllin, nitroglycerine) or anticoagulating drugs (e.g. heparine, cumarines, new oral anticoagulants, regular intake of acetylsalicylic acid)
21. Current or within 3 months prior to first dosing use of systemic corticosteroids (nose drops, eye drops and/or inhalers are permitted) or other immunosuppressive drugs (e.g. cyclosporine A)
22. Elevated values for vital signs: blood pressure: systolic above 160 mmHg, diastolic above 95 mmHg, pulse rate: above 100 beats/min
23. Planned or scheduled subject surgery or hospitalisation during the course of the trial
24. Previously randomized in this trial (only valid for subjects included after 01JUN2020)
25. Psychiatric conditions that might limit the participation in the trial and/or that lead to the assumption that the ability to completely understand the consequences of consent is missing.
26. Subjects, who are inmates of psychiatric wards, prisons or state institutions.
27. Participation in a clinical trial with investigational medicinal products within the last 30 days prior to the Day 1 and / or during this trial.
28. Employees of the trial sites who are directly involved in this trial or employees of the Sponsor's company.
29. If in the opinion of the Investigator the subject should not participate in the trial for any reason.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

PRIMARY OUTCOMES:
Change in total hair density at week 16 | 16 weeks
  The change in total (terminal+vellus) hair density (hair count (n per cm²)) from Baseline to Day 112

SECONDARY OUTCOMES:
Change in total hair density at week 12 | 12 weeks
  The change in total (terminal+vellus) hair density (hair count (n per cm²)) from Baseline to Day 84
Change in terminal hair density at week 16 | 16 week
  Comparisons of treatments on terminal hair density at week 16 based on relative differences to Baseline
Change in vellus hair density at week 16 | 16 week
  Comparisons of treatments on vellus hair density at week 16 based on relative differences to Baseline
Change in telogen hair density at week 16 | 16 weeks
  Comparison of the change from Baseline (Day 1) to week 16 in percentage of telogen hairs (number of telogen hairs /total number of hairs) for each IP separately
Change in anagen hair density at week 16 | 16 weeks
  Comparison of the change from Baseline (Day 1) to week 16 in percentage of anagen hairs (number of anagen hairs /total number of hairs) for each IP separately
Safety parameters | 16 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Blume-Peytavi, Principal Investigator — Klinik für Dermatologie, Charité-Universitätsmedizin, Berlin
Locations (1):
- ProDerm GmbH, Hamburg, Germany